CLINICAL TRIAL: NCT06210334
Title: The Safety and Efficacy of Hepatic Arterial Infusion Chemotherapy (HAIC) Combine Tislelizumab and Lenvatinib in the Treatment of Hepatocellular Carcinoma (HCC) With Type IV(Vp4) Portal Vein Tumor Thrombus (PVTT): A Prospective, Single-armed, Stage II Clinical Trial
Brief Title: HAIC Combine Tislelizumab and Lenvatinib in the Treatment of HCC With Type IV (Vp4) Portal Vein Tumor Thrombus (HAI-TL)
Acronym: HAI-TL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Li Xiao Wei (Other)
Responsible Party: Sponsor-Investigator, Li Xiao Wei, Associate chief physician, Eastern Hepatobiliary Surgery Hospital
Organization: Eastern Hepatobiliary Surgery Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EasternHSH-IR
Record Dates: First submitted 2024-01-02; First posted 2024-01-18 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Hepatocellular Carcinoma With PVTT
Keywords: Hepatocellular Carcinoma; Hepatic Arterial Infusion Chemotherapy; Portal Vein Tumor Thrombus; Tislelizumab; Lenvatinib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tislelizumab; lenvatinib

STUDY DESIGN:
Intervention Model Description: A Prospective, Single-armed, Stage II Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC combined with Tislelizumab and Lenvatinib (HAI-TIS-LEN) group (Experimental): HAIC with modified FOLFOX (oxaliplatin, 85 mg/ m2, leucovorin 400 mg/ m2, 5-fluorouracil bolus 400 mg/m2 on day 1; and 5-fluorouracil infusion 2400 mg/ m2 for 46 h) on day1-2 every 3 weeks. Tislelizumab injection intravenously after 24h of HAIC every 3 week. Lenvatinib 12/8 mg (weight ≥ 60 kg/< 60 kg) orally once daily starting 1-3 days after HAIC.
  Interventions: Drug: Tislelizumab; Drug: Lenvatinib

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200mg, iv, d3, q3w
  Other Names: PD-1
Drug: Lenvatinib — Lenvatinib 8mg (<60kg) or 12mg (≥60kg), po, qd
  Other Names: TKI

SUMMARY:
To estimate the safety and efficacy of hepatic artery infusion chemotherapy (HAIC) combine Tislelizumab and Lenvatinib (HAI-TIS-LEN) in the Treatment of hepatocellular carcinoma (HCC) with type IV(Vp4) portal vein tumor thrombus (PVTT).

DETAILED DESCRIPTION:
According to the Chinese guidelines for the diagnosis and treatment of primary liver cancer, patients with hepatocellular carcinoma (HCC) accompanied by portal vein tumor thrombosis (PVTT) are classified as being in an advanced stage (CNLC IIIa). PVTT, particularly the type IV (Vp4), is considered a highly concerning complication of HCC due to its significant morbidity and mortality rates. Furthermore, the absence of effective treatment options contributes to an unfavorable prognosis.

Hepatic arterial infusion chemotherapy (HAIC) delivers chemotherapy drugs directly through a catheter into the nourishing arteries of the tumor, maintaining a high concentration of chemotherapeutic agents within the tumor and tumor thrombus, thereby promoting necrosis. HAIC with modified FOLFOX (oxaliplatin, 85 mg/m2, leucovorin 400 mg/m2, 5-fluorouracil bolus 400 mg/m2 on day 1; and 5-fluorouracil infusion 2400 mg/m2 for 46 h) could significantly prolong survival time for HCC patients with PVTT.

In recent years, official guidelines have approved several immune checkpoint inhibitors for advanced HCC. Lenvatinib, an innovative oral anti-neovascularity inhibitor, has demonstrated comparable efficacy to sorafenib in HCC patients, as evidenced by the REFLECT study. Additionally, the exploration of programmed death-1 (PD-1) inhibitors, either alone or in combination with targeted therapy, has been confirmed as effective for advanced HCC.

Against this background, researchers have initiated a prospective, single-arm, Stage II clinical trial to assess the effectiveness and safety of HAIC combined with Tislelizumab and Lenvatinib (HAI-TIS-LEN) for advanced HCC with Vp4 involvement. A total of 45 subjects will be enrolled in this trial. The primary endpoint of the study is the median overall survival (mOS), the secondary endpoints including the overall response rate (ORR), disease control rate (DCR), median progression-free survival (mPFS), time-to-progression (TTP), and safety assessment. The safety assessment will be conducted in accordance with the standard adverse reaction classification outlined in the Common Terminology Criteria for Adverse Events (CTCAE v5.0).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically, cytologically, or clinically confirmed diagnosis of hepatocellular carcinoma (HCC).
2. Age between 18 and 75 years.
3. Presence of type 4 portal vein tumor thrombosis (PVTT).
4. Child-Pugh A or B liver function.
5. Eastern Cooperative Group performance status (ECOG) score of 0-2.
6. Satisfactory blood, liver, and kidney function parameters, including:

   * (a) Hemoglobin concentration ≥ 8.5 g/dL, neutrophil count ≥ 1.5 × 10^9/L, platelet count ≥ 40 × 10^9/L.
   * (b) Serum albumin concentration ≥ 30 g/L, bilirubin ≤ 50 μmol/L, AST and ALT < 5 × upper limit of normal (ULN), and alkaline phosphatase < 4 × ULN.
   * (c) Extended prothrombin time < 6 seconds of ULN.
   * (d) Serum creatinine < 1.5 × ULN.
7. Ability to comprehend the protocol and provide informed consent by signing a written document.

Exclusion Criteria:

1. History of a second primary malignant tumor.
2. Severe dysfunction of the heart, kidneys, or other organs.
3. Evidence of hepatic decompensation, including ascites, active gastrointestinal bleeding, or hepatic encephalopathy.
4. Pregnancy or lactation.
5. Known history of HIV.
6. History of organ allograft.
7. Known or suspected allergy to investigational agents or any agent administered in conjunction with this trial.
8. Active gastric or duodenal ulcers within 3 months before enrollment.
9. Incomplete medical data or loss to follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From the date of treatment initiation until the date of death from any cause, assessed up to 60 months.
  Duration from the date of initial HAI-TIS-LEN treatment to the date of death due to any cause.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | The average expectation is 36 months.
  Defined as the time from the treatment initiation to the date of the first objectively documented tumor progression or death, whichever occurs first, assessed by IRC and investigators, respectively, per RECIST v 1.1 and mRECIST.
Time-to-progression (TTP) | The average expectation is 36 months.
  Defined as the time from treatment initiation to radiological progression.
Objective Response Rate (ORR) | On average once every month, assessed up to 36 months.
  Defined as the proportion of participants in the study population who achieve a complete response (CR) or partial response (PR), as determined by investigators using the RECIST v 1.1 and mRECIST criteria, at any time during the study.
Disease Control Rate (DCR) | On average once every month, assessed up to 36 months.
  Defined as the proportion of patients whose best overall response is CR, PR, or SD, assessed by investigators, per RECIST v 1.1 and mRECIST
Adverse Events (AE) | From the date of treatment initiation until 60 days after the last treatment.
  Any adverse events related to treatment drugs, including details such as adverse event type, frequency, and severity.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhai, MM, Study Director — Eastern Hepatobiliary Surgery Hospital
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Yangpu, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be openly available in Research Data Deposit at https://www.researchdata.org.cn, after publication.
Supporting Information: CSR
Time Frame: Submission of data starting 6 months after publication, expected to be open for 6 months.
Access Criteria: open
URL: https://www.researchdata.org.cn/

REFERENCES:
- [Background] Zhou J, Sun H, Wang Z, Cong W, Zeng M, Zhou W, Bie P, Liu L, Wen T, Kuang M, Han G, Yan Z, Wang M, Liu R, Lu L, Ren Z, Zeng Z, Liang P, Liang C, Chen M, Yan F, Wang W, Hou J, Ji Y, Yun J, Bai X, Cai D, Chen W, Chen Y, Cheng W, Cheng S, Dai C, Guo W, Guo Y, Hua B, Huang X, Jia W, Li Q, Li T, Li X, Li Y, Li Y, Liang J, Ling C, Liu T, Liu X, Lu S, Lv G, Mao Y, Meng Z, Peng T, Ren W, Shi H, Shi G, Shi M, Song T, Tao K, Wang J, Wang K, Wang L, Wang W, Wang X, Wang Z, Xiang B, Xing B, Xu J, Yang J, Yang J, Yang Y, Yang Y, Ye S, Yin Z, Zeng Y, Zhang B, Zhang B, Zhang L, Zhang S, Zhang T, Zhang Y, Zhao M, Zhao Y, Zheng H, Zhou L, Zhu J, Zhu K, Liu R, Shi Y, Xiao Y, Zhang L, Yang C, Wu Z, Dai Z, Chen M, Cai J, Wang W, Cai X, Li Q, Shen F, Qin S, Teng G, Dong J, Fan J. Guidelines for the Diagnosis and Treatment of Primary Liver Cancer (2022 Edition). Liver Cancer. 2023 Apr 5;12(5):405-444. doi: 10.1159/000530495. eCollection 2023 Oct. PMID 37901768
- [Background] Thomas MB, Jaffe D, Choti MM, Belghiti J, Curley S, Fong Y, Gores G, Kerlan R, Merle P, O'Neil B, Poon R, Schwartz L, Tepper J, Yao F, Haller D, Mooney M, Venook A. Hepatocellular carcinoma: consensus recommendations of the National Cancer Institute Clinical Trials Planning Meeting. J Clin Oncol. 2010 Sep 1;28(25):3994-4005. doi: 10.1200/JCO.2010.28.7805. Epub 2010 Aug 2. PMID 20679622
- [Background] Finn RS, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Xu DZ, Hernandez S, Liu J, Huang C, Mulla S, Wang Y, Lim HY, Zhu AX, Cheng AL; IMbrave150 Investigators. Atezolizumab plus Bevacizumab in Unresectable Hepatocellular Carcinoma. N Engl J Med. 2020 May 14;382(20):1894-1905. doi: 10.1056/NEJMoa1915745. PMID 32402160
- [Background] Ren Z, Xu J, Bai Y, Xu A, Cang S, Du C, Li Q, Lu Y, Chen Y, Guo Y, Chen Z, Liu B, Jia W, Wu J, Wang J, Shao G, Zhang B, Shan Y, Meng Z, Wu J, Gu S, Yang W, Liu C, Shi X, Gao Z, Yin T, Cui J, Huang M, Xing B, Mao Y, Teng G, Qin Y, Wang J, Xia F, Yin G, Yang Y, Chen M, Wang Y, Zhou H, Fan J; ORIENT-32 study group. Sintilimab plus a bevacizumab biosimilar (IBI305) versus sorafenib in unresectable hepatocellular carcinoma (ORIENT-32): a randomised, open-label, phase 2-3 study. Lancet Oncol. 2021 Jul;22(7):977-990. doi: 10.1016/S1470-2045(21)00252-7. Epub 2021 Jun 15. PMID 34143971
- [Background] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Background] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- Available data/document: Clinical Study Report — https://www.researchdata.org.cn/